CLINICAL TRIAL: NCT03640728
Title: A Multicenter Controlled Open-label Trial of Evaluating Tenofovir Alafenamide, Tenofovir Disoproxil Fumarate and Entecavir in Acute-on-chronic Liver Failure of Chronic Hepatitis B Patients
Brief Title: The Efficacy and Safety of Nucleos(t)Ide Analogues in the Treatment of HBV-related Acute-on-chronic Liver Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, He Yingli, He Yingli, Research Associate, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: XJTU1AF2018LSL-002
Record Dates: First submitted 2018-08-19; First posted 2018-08-21 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Hepatitis B; Virus Diseases; Liver Failure
Keywords: Hepatitis B, Acute-on-Chronic liver failure
MeSH Terms: conditions — Hepatitis B; Virus Diseases; Liver Failure; Acute-On-Chronic Liver Failure | interventions — tenofovir alafenamide; entecavir; Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ETV: patients receive entecavir 0.5 mg/day orally.
  Interventions: Drug: Entecavir
- TDF: patients receive Tenofovir Disoproxil Fumarate 300 mg/day orally.
  Interventions: Drug: Tenofovir disoproxil fumarate
- TAF: patients receive Tenofovir alafenamide 25 mg/day orally.
  Interventions: Drug: Tenofovir Alafenamide

INTERVENTIONS:
Drug: Tenofovir Alafenamide — Tenofovir alafenamide 25 mg/day orally
  Groups: TAF
Drug: Entecavir — Entecavir 0.5 mg/day orally
  Groups: ETV
Drug: Tenofovir disoproxil fumarate — Tenofovir Disoproxil Fumarate 300 mg/day orally
  Groups: TDF

SUMMARY:
HBV-related acute-on-chronic liver failure (ACLF) is a clinical syndrome defined as acute hepatic insult with diagnosed or undiagnosed chronic liver disease. Current clinical guidelines advocate oral antiviral treatment in HBV-related ACLF. However, no conclusion on which nucleoside analogue is the most satisfactory drug for the treatment of HBV-related liver failure has not been reached yet. In this cohort study, the investigators will compare the efficacy, safety, and tolerability of tenofovir alafenamide (TAF), Tenofovir Disoproxil Fumarate (TDF) and entecavir (ETV) in HBV-related ACLF in China. In addition, the drug metabolism characteristics of TAF will be explored in such severe liver injury population of HBV-ACLF.

DETAILED DESCRIPTION:
Potent antivirals like entecavir (ETV), Tenofovir Disoproxil Fumarate (TDF) and Tenofovir alafenamide (TAF) now are recommended as first-line therapy for patients with chronic HBV infection because of their significant suppression of viral replication and a high barrier to resistance. HBV-related acute-on-chronic liver failure (ACLF) is a clinical syndrome defined as acute hepatic insult with diagnosed or undiagnosed chronic liver disease. Only a limited number of medical treatments are available for ACLF. Although liver transplantation is a life-saving treatment for ACLF, the difficulty in finding a suitable donor and the high cost hinder its extensive clinical use.

The precise mechanism underlying the liver injury caused by HBV-related ACLF and the factors contributing to the progression of liver failure remain unknown. HBV DNA replication is one of the key factors causing the progression from liver damage to liver failure. Current clinical guidelines advocate oral antiviral treatment in HBV-related ACLF. However, the specific antiviral treatment for patients with liver failure remains unclear. In the past years, efficacy of nucleoside analogues, such as lamivudine, entecavir, telbivudine and tenofovir, for HBV-related liver failure has been reported. However, no conclusion on which nucleoside analogue is the most satisfactory drug for the treatment of HBV-related liver failure has not been reached yet.

In this cohort study, the investigators will compare the efficacy, safety, and tolerability of tenofovir alafenamide (TAF), Tenofovir Disoproxil Fumarate (TDF) and entecavir (ETV) in HBV-related ACLF in China. In addition, pharmacokinetic properties of TAF tablets will be explored in the study subjects.

ELIGIBILITY:
Inclusion Criteria:All of below

1. age 18-70 years, male or female.
2. HBsAg positive at least 6 months or more, HBeAg positive or negative.
3. Serum HBV DNA positive (Serum HBV DNA should be determined by the PCR assay at the local laboratory at screening for this study)
4. Recent development of increasing jaundice (a total serum bilirubin concentration of above 85μmol/L) and coagulopathy (INR ≥1.5 or prothrombin activity<40%)
5. Recent development of complications such as hepatic encephalopathy, or abrupt and obvious increase in ascites, or spontaneous bacterial peritonitis, or hepatorenal syndrome.
6. Patient is willing and able to comply with the study drug regimen and all other study requirements.
7. The patient is willing and able to provide written informed consent to participate in the study.

Exclusion Criteria: Any of below

1. Patient has concomitant other chronic viral infection (HCV or HIV)
2. Patient has evidence of renal insufficiency defined as serum creatinine > 1.5 mg/dL
3. Patient has medical condition that requires concurrent use of systemic prednisolone or other immunosuppressive agent (including chemotherapeutic agent)
4. Patient is pregnant or breastfeeding or willing to be pregnant
5. Patient has one or more additional known primary or secondary causes of liver disease, other than hepatitis B (e.g., alcoholism, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's Disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease, etc.).
6. A history of treated malignancy (other than hepatocellular carcinoma) is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding three years.
7. Active ethanol/drug abuse/psychiatric problems such as major depression, schizophrenia, bipolar illness, obsessive-compulsive disorder, severe anxiety, personality disorder that might interfere with participation in the study.
8. Current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients received antivirals will be followed for at least 48 weeks and follow-up assessments were performed at week 1, 2, 3, 4, 12, 24 and 48.All the patients were detected Serum HBV DNA,HBV markers, including HBsAg, HBsAb, HBeAg, HBeAb and HBcAb, routine biochemical tests mainly including ALT,AST,TB and ALB.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival of ACLF subjects | study day 1 through week 48
  Overall survival in subjects with acute-on-chronic liver failure will be summarized and compared with control subjects through study day 28 and week 48.

SECONDARY OUTCOMES:
Changes in serum HBV DNA levels | at week 4 and 48 of treatment
Proportion of patients with hepatitis B e-Ag(HBe-Ag) loss or seroconversion | at week 4 and 48 of treatment
Proportion of patients with HBs-Ag loss or seroconversion | at week 4 and 48 of treatment
Proportion of patients with normal alanine aminotransferase(ALT) | at week 4 and 48 of treatment
Liver function evaluation through Model for End-Stage Liver Disease (MELD) scores | at week 4 and 48 of treatment
  Model for End-Stage Liver Disease(MELD) Score is calculated according to the equation:3.78×ln[serum bilirubin (mg/dl)] + 11.2×ln(INR) + 9.57×ln[serum creatinine (mg/dL)] + 6.43. Liver function improvement defined as the decline of total MELD score, whereas liver function deterioration defined as the rise of total MELD score. The risk of death increased when total MELD score above 25.
Proportion of patients with virologic breakthrough | at week 4 and 48 of treatment
  Virologic breakthrough is defined as the increase in serum HBV DNA by >1 log10 (10-fold) above nadir after achieving virologic response as determined by at least 2 consecutive measurements of at least 2 weeks apart, during continued treatment
Proportion of patients with complete virologic response | at week 4 and 48 of treatment
  Virologic response is defined as the serum HBV DNA concentrations below 20 IU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Yingli He, M.D.,Ph.D, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (11):
- China (11):
  - Ankang Central Hospital, Ankang
  - Hanzhong 3201 Hospital, Hanzhong
  - Hanzhong Infectious Hospital, Hanzhong
  - Weinan Central Hospital, Weinan
  - First Affiliated Hospital Xi'an Jiaotong University, Xi'an
  - Shaanxi provincial people's hospital, Xi'an
  - Tangdu Hospital, The Fourth Military Medical University,, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xi'an Central Hospital, Xi'an
  - Xijing Hospital, The Fourth Military Medical University, Xi'an
  - The Affiliated Hospital of Yan'an University, Yan’an

REFERENCES:
- [Derived] Li J, Hu C, Chen Y, Zhang R, Fu S, Zhou M, Gao Z, Fu M, Yan T, Yang Y, Li J, Liu J, Chen T, Zhao Y, He Y. Short-term and long-term safety and efficacy of tenofovir alafenamide, tenofovir disoproxil fumarate and entecavir treatment of acute-on-chronic liver failure associated with hepatitis B. BMC Infect Dis. 2021 Jun 14;21(1):567. doi: 10.1186/s12879-021-06237-x. PMID 34126939